CLINICAL TRIAL: NCT05468398
Title: The Effect of Virtual Reality on Pain and Patient Satisfaction in Adults Receiving Genicular Nerve Radiofrequency Ablation
Brief Title: Effect of VR on Pain and Patient Satisfaction in Adults Receiving GNRFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Applied VR (Unknown)
Responsible Party: Principal Investigator, Navid Alem, Associate Clinical Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20206207
Record Dates: First submitted 2022-02-18; First posted 2022-07-21 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Pain; Patient Satisfaction
Keywords: Genicular Nerve Block; Virtual Reality; Genicular Nerve Radiofrequency Ablation; GNRFA
MeSH Terms: conditions — Pain; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This was a single-center, non-blinded, randomized controlled trial with a parallel assignment design. Participants were randomly allocated in a 1:1 ratio to receive either standard care alone or standard care with immersive virtual reality (VR) therapy during genicular nerve radiofrequency ablation (GNRFA). The intervention was administered during the procedure only. The study aimed to assess the impact of VR on patient-reported pain, anxiety, satisfaction, and physician-rated procedural outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): The control group will receive a genicular RFA with local anesthetic as per the standard-of-care
- VR Intervention (Experimental): The VR Intervention group will receive a genicular RFA with local anesthetic as per the standard-of-care and the use of the Soothe VR device.
  Interventions: Device: Soothe VR

INTERVENTIONS:
Device: Soothe VR — The Soothe VR system is manufactured by Applied VR. It is a HIPAA-compliant platform and has been validated by randomized control trials. It has not yet been reviewed by the FDA.
  Arms: VR Intervention

SUMMARY:
The study team aims to investigate whether implementing virtual reality therapy (VRT) during Genicular nerve radiofrequency ablation (GNRFA) procedure will provide better alleviation of procedural pain and augmented satisfaction for patients.

DETAILED DESCRIPTION:
Patients' experience through a medical procedure in a hospital environment is inherently stressful and painful. Although virtual reality (VR) was originally recognized for its entertainment value, it has recently been used as an innovative tool in clinical settings to reduce pain and anxiety, while improving patient satisfaction. VR is a computer generated simulation of a life-like experience that usually serves people for entertainment and social interactive purposes in a simulated three-dimensional environment. Virtual reality therapy (VRT) offers patients an opportunity to "get away" from noxious stimuli as they draw their attention towards another virtual world (Alem).

Virtual reality provides a cognitive distraction through creating a "real world illusion." VR may deter an individual's attention from pain as it offers a multimodal sensory distractor. This positive experience may result in reduction of pain score by decreasing the time patients think about their pain during a procedure.

Genicular nerve radiofrequency ablation (GNRFA) is an option to treat knee pain without surgery. The genicular nerves are the nerves that feed into the knee. Radiofrequency ablation is a process by applying radiofrequency waves to the nerves that are carrying the painful impulses from the knee joint. GNRFA uses fluoroscopy guidance to introduce 3 needles at each of the three genicular nerves which transmit sensation from the knee joint. This is followed by testing for sensory response, followed by administration of local anesthetic (2% lidocaine) per standard-of-care, and then radiofrequency ablation. This method of treatment is known to be very safe, convenient and reliable because fluoroscopy guidance provides high accuracy of localization at the procedure targets outside of the knee joint. Patients with symptomatic knee osteoarthritis have shown short and long term positive results following this method with significant reduction of pain levels (Kidd) and augmented functionality. This non-invasive procedure is able to successfully replace surgery or intra-articular therapy where the procedure is conducted directly on the knee joint.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 or older
* Patients Undergoing a genicular nerve radiofrequency ablation
* Patients who have previously received nerve blocks or radiofrequency ablation procedures may be included

Exclusion Criteria:

* Requiring sedation during procedure
* Cognitive impairment or dementia
* History of recent stroke, epilepsy, psychosis, or claustrophobia
* Blindness or deafness
* Refusal to use the headset
* Isolation status for infection control
* Motion sickness or active nausea/vomit
* Pregnancy (Pregnancy testing point of care available for females of child bearing age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Navid Alem, MD, Principal Investigator — Faculty
Locations (1):
- UC Irvine Gottschalk Medical Plaza, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alaterre C, Duceau B, Sung Tsai E, Zriouel S, Bonnet F, Lescot T, Verdonk F. Virtual Reality for PEripheral Regional Anesthesia (VR-PERLA Study). J Clin Med. 2020 Jan 13;9(1):215. doi: 10.3390/jcm9010215. PMID 31941129
- [Background] Kidd VD, Strum SR, Strum DS, Shah J. Genicular Nerve Radiofrequency Ablation for Painful Knee Arthritis: The Why and the How. JBJS Essent Surg Tech. 2019 Mar 13;9(1):e10. doi: 10.2106/JBJS.ST.18.00016. eCollection 2019 Mar 26. PMID 31333900
- [Background] Jamison DE, Cohen SP. Radiofrequency techniques to treat chronic knee pain: a comprehensive review of anatomy, effectiveness, treatment parameters, and patient selection. J Pain Res. 2018 Sep 18;11:1879-1888. doi: 10.2147/JPR.S144633. eCollection 2018. PMID 30271194
- [Background] Hong T, Wang H, Li G, Yao P, Ding Y. Systematic Review and Meta-Analysis of 12 Randomized Controlled Trials Evaluating the Efficacy of Invasive Radiofrequency Treatment for Knee Pain and Function. Biomed Res Int. 2019 Jun 26;2019:9037510. doi: 10.1155/2019/9037510. eCollection 2019. PMID 31346525
- [Background] Chan PY, Scharf S. Virtual Reality as an Adjunctive Nonpharmacological Sedative During Orthopedic Surgery Under Regional Anesthesia: A Pilot and Feasibility Study. Anesth Analg. 2017 Oct;125(4):1200-1202. doi: 10.1213/ANE.0000000000002169. PMID 28598921
- [Background] McCaul KD, Malott JM. Distraction and coping with pain. Psychol Bull. 1984 May;95(3):516-33. No abstract available. PMID 6399756
- [Background] Mahrer NE, Gold JI. The use of virtual reality for pain control: a review. Curr Pain Headache Rep. 2009 Apr;13(2):100-9. doi: 10.1007/s11916-009-0019-8. PMID 19272275
- [Background] Hoffman HG, Seibel EJ, Richards TL, Furness TA, Patterson DR, Sharar SR. Virtual reality helmet display quality influences the magnitude of virtual reality analgesia. J Pain. 2006 Nov;7(11):843-50. doi: 10.1016/j.jpain.2006.04.006. PMID 17074626
- [Background] Mosso JL, Gorini A, De La Cerda G, Obrador T, Almazan A, Mosso D, Nieto JJ, Riva G. Virtual reality on mobile phones to reduce anxiety in outpatient surgery. Stud Health Technol Inform. 2009;142:195-200. PMID 19377147
- [Background] Carrougher GJ, Hoffman HG, Nakamura D, Lezotte D, Soltani M, Leahy L, Engrav LH, Patterson DR. The effect of virtual reality on pain and range of motion in adults with burn injuries. J Burn Care Res. 2009 Sep-Oct;30(5):785-91. doi: 10.1097/BCR.0b013e3181b485d3. PMID 19692911
- [Background] Sharar SR, Carrougher GJ, Nakamura D, Hoffman HG, Blough DK, Patterson DR. Factors influencing the efficacy of virtual reality distraction analgesia during postburn physical therapy: preliminary results from 3 ongoing studies. Arch Phys Med Rehabil. 2007 Dec;88(12 Suppl 2):S43-9. doi: 10.1016/j.apmr.2007.09.004. PMID 18036981
- [Background] Spiegel B, Fuller G, Lopez M, Dupuy T, Noah B, Howard A, Albert M, Tashjian V, Lam R, Ahn J, Dailey F, Rosen BT, Vrahas M, Little M, Garlich J, Dzubur E, IsHak W, Danovitch I. Virtual reality for management of pain in hospitalized patients: A randomized comparative effectiveness trial. PLoS One. 2019 Aug 14;14(8):e0219115. doi: 10.1371/journal.pone.0219115. eCollection 2019. PMID 31412029
- [Background] Sikka N, Shu L, Ritchie B, Amdur RL, Pourmand A. Virtual Reality-Assisted Pain, Anxiety, and Anger Management in the Emergency Department. Telemed J E Health. 2019 Dec;25(12):1207-1215. doi: 10.1089/tmj.2018.0273. Epub 2019 Feb 20. PMID 30785860
- [Background] Gold JI, Mahrer NE. Is Virtual Reality Ready for Prime Time in the Medical Space? A Randomized Control Trial of Pediatric Virtual Reality for Acute Procedural Pain Management. J Pediatr Psychol. 2018 Apr 1;43(3):266-275. doi: 10.1093/jpepsy/jsx129. PMID 29053848
- See also: Applied VR Research Studies — https://www.appliedvr.io/research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at University of California, Irvine Health's Gottschalk Medical Plaza between December 2020 and September 2024. Due to study scope and completion of planned enrollment, the study closed with 40 enrolled participants.
Pre-assignment Details: Of the 40 participants who consented, all were randomized.
Period: Overall Study
Arm/Group | Control | VR Intervention
Started | 18 | 22
Completed | 18 | 21
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: All 40 participants (22 in the VR group, 18 in the control group) completed baseline surveys and were included in the baseline analysis. Each participant contributed one unit of analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | VR Intervention | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.4) | 65.2 (8.7) | 65.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 22 | 40
Baseline pain intensity was measured using the Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale 0 - 100] — The VAS assesses the participant's perceived pain level on a continuous scale ranging from 0 (no pain) to 100 (worst imaginable pain). Higher scores indicate worse pain.
  units on a scale 0 - 100 | 66.3 (9.4) | 65.2 (8.7) | 65.7 (9.0)

OUTCOME MEASURES:

1. Primary Outcome: Peak Pain Intensity During Genicular RFA Procedure
Description: Peak pain intensity experienced by participants during the genicular RFA procedure was assessed using a Graphic Rating Scale (GRS) from 0 (no pain) to 100 (worst imaginable pain). Higher scores indicate greater pain intensity (worse outcome).
Time Frame: 20 minutes
Population: All participants who completed both the pre- and post-procedure pain assessments were included in this analysis (n=40). Pain score reduction was calculated as the difference between pre- and post-procedure VAS scores.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control | VR Intervention
Number analyzed (Participants) | 18 | 22
units on a scale | 78.17 (18.25) | 68.17 (24)

2. Primary Outcome: Patient Satisfaction With VR Device
Description: Patient satisfaction with the Virtual Reality (VR) device during the genicular radiofrequency ablation (RFA) procedure was assessed using a Graphic Rating Scale (GRS). Participants rated their overall satisfaction immediately following the procedure on a continuous scale ranging from 0 (not satisfied at all) to 100 (extremely satisfied). Higher scores indicate greater satisfaction, representing a better outcome.
Time Frame: Immediately post-genicular RFA procedure (approximately 20 minutes after procedure initiation)
Population: Only participants in the VR group completed the satisfaction survey. All 22 participants in this group were included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a 0 -100 scale
Arm/Group | VR Intervention
Number analyzed (Participants) | 22
units on a 0 -100 scale | 87.7 (15.6)

3. Secondary Outcome: Duration of Time Patient Spent Thinking About Pain During Genicular RFA Procedure
Description: The duration or proportion of time patients spent thinking about their pain during the genicular radiofrequency ablation (RFA) procedure was assessed using a 0-100 Graphic Rating Scale (GRS). Participants rated how much time they spent thinking about pain during the procedure, with scores ranging from 0 ("no time thinking about pain") to 100 ("entire procedure spent thinking about pain"). Higher scores indicate a worse outcome (greater proportion of procedure time spent thinking about pain).
Time Frame: During the genicular RFA procedure (approximately 20 minutes)
Reporting Status: Not Posted

4. Secondary Outcome: Patient Anxiety During Genicular RFA Procedure Patient Anxiety During Genicular RFA Procedure Patient Anxiety During Genicular RFA Procedure
Description: Patient anxiety during the genicular radiofrequency ablation (RFA) procedure was assessed using a 0-100 Graphic Rating Scale (GRS). Patients rated their anxiety level during the procedure only, from 0 ("not anxious at all") to 100 ("extremely anxious"). Higher scores indicate a worse outcome (greater anxiety).
Time Frame: During the genicular RFA procedure (approximately 20 minutes)
Population: All 40 participants (22 in the VR group, 18 in the control group) completed the anxiety question during the procedure and were included in this analysis. Anxiety was measured using a 0-100 Graphic Rating Scale, with higher scores indicating greater anxiety.
Measure: Mean (Standard Deviation); unit: Units on a 0-100 scale
Arm/Group | Control | VR Intervention
Number analyzed (Participants) | 18 | 22
Units on a 0-100 scale | 71.17 (23.15) | 51.4 (26.13)

5. Secondary Outcome: Provider Satisfaction During Procedure
Description: Practitioners' satisfaction with the Virtual Reality (VR) device during the genicular radiofrequency ablation (RFA) procedure was assessed using a 0-100 Graphic Rating Scale (GRS). Providers rated their overall satisfaction immediately following completion of the procedure, from 0 ("not satisfied at all") to 100 ("extremely satisfied"). Higher scores indicate greater satisfaction, representing a better outcome.
Time Frame: Immediately post-genicular RFA procedure (approximately 20 minutes after procedure initiation)
Population: Practitioners rated their satisfaction with the procedure using a 0-100 Graphic Rating Scale. Higher scores indicate greater satisfaction. Surveys were completed after each procedure based on the provider's experience with patient behavior and ease of the procedure.
Measure: Mean (Standard Deviation); unit: Units on a 0-100 scale
Arm/Group | Control | VR Intervention
Number analyzed (Participants) | 18 | 22
Units on a 0-100 scale | 61.25 (24) | 87.9 (15.25)

6. Secondary Outcome: Use of Additional Local Anesthetic During Genicular RFA Procedure
Description: The need for additional local anesthetic administration during the genicular radiofrequency ablation (RFA) procedure was assessed as a binary outcome (Yes/No). Providers recorded whether additional local anesthetic was administered beyond the standard initial dose during the procedure.
Time Frame: During the genicular RFA procedure (approximately 20 minutes)
Reporting Status: Not Posted

7. Secondary Outcome: Provider Perception of Patient's Pain During Genicular RFA Procedure
Description: Provider's perception of the patient's pain during the genicular RFA procedure was assessed using a 0-100 Graphic Rating Scale (GRS). Providers rated their perception of patient pain from 0 ("no perceived pain") to 100 ("extremely severe pain"). Higher scores indicate a worse outcome (higher perceived patient pain).
Time Frame: During the genicular RFA procedure (approximately 20 minutes)
Population: Ratings were based on provider observation and recorded using a 0-100 Graphic rating Scale, where higher scores indicate greater perceived patient pain.
Measure: Mean (Standard Deviation); unit: Units on a 0-100 Scale
Arm/Group | Control | VR Intervention
Number analyzed (Participants) | 18 | 22
Units on a 0-100 Scale | 71.11 (18.50) | 36.74 (21.67)

8. Secondary Outcome: Prior Knee Radiofrequency Ablation
Description: Participants were asked if they had undergone a previous knee radiofrequency ablation (RFA) procedure prior to the study intervention. Responses were recorded as binary outcomes (Yes/No).
Time Frame: Assessed at baseline (participant history of knee RFA within the past 2 years)
Reporting Status: Not Posted

9. Secondary Outcome: Prior Experience With Virtual Reality (VR)
Description: Participants reported if they had previously used Virtual Reality (VR) technology for any reason (e.g., gaming, therapy) before participation in the study. Responses were recorded as binary outcomes (Yes/No).
Time Frame: Assessed at baseline (participant history of VR use within the past 2 years)
Reporting Status: Not Posted

10. Secondary Outcome: Side Effects Associated With Virtual Reality During Genicular RFA Procedure
Description: Participants were asked immediately after the procedure if they experienced any side effects related to the use of Virtual Reality (VR), such as headache, dizziness, nausea, or palpitations. Responses were recorded as binary outcomes (Yes/No).
Time Frame: Immediately post-procedure (approximately 20 minutes after procedure initiation)
Reporting Status: Not Posted

11. Secondary Outcome: Subgroup Analysis by Age, Gender, Provider, and Technology Acceptance
Description: A descriptive subgroup analysis of participants was conducted to identify commonalities in response and acceptance of technology across demographic characteristics including age, gender, provider type, and general acceptance of technology.
Time Frame: Assessed at baseline (demographic information collected at enrollment)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Participants were monitored continuously during and immediately following the genicular RFA procedure (approximately 20 minutes after procedure initiation).
Description: Participants were continuously observed by clinical personnel for any adverse events (serious or non-serious) during and immediately following the genicular RFA procedure.
Arm/Group | Control | VR Intervention
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/22
Other Adverse Events (participants affected / at risk) | 0/18 | 0/22

LIMITATIONS AND CAVEATS:
This was a single-site, randomized but non-blinded pilot study with a relatively small sample size, which may limit generalizability. Participants and providers were aware of group assignments when the VR device was applied. Self-reported measures and a study pause due to COVID-19 may have impacted data consistency.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-23): https://cdn.clinicaltrials.gov/large-docs/98/NCT05468398/Prot_SAP_003.pdf
  • Informed Consent Form (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT05468398/ICF_001.pdf